CLINICAL TRIAL: NCT03683602
Title: Effect of Chosen Treatment Methods on Pain, ROM, Associated Symptoms and Functioning in Patients With Cervical Spine Osteoarthritis: Randomised Control Trial
Brief Title: Effect of Chosen Treatment Methods in Patients With Cervical Spine Osteoarthritis
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Maicki, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NECK/2018
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Cervical Spine Osteophyte
Keywords: PNF, manual therapy, neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF group (Experimental): PNF techniques, patterns, re-education of postural control, once a day 10 days,
  Interventions: Other: PNF group
- Manual therapy group (Active Comparator): traction, joints mobilization, pos-isometric relaxation, once a day 10 days
  Interventions: Other: manual therapy group

INTERVENTIONS:
Other: PNF group — PNF is used in treatment of musculoskeletal pain of cervical and lumbar spine. Proprioceptive neuromuscular facilitation is a rehabilitation concept widely used by physiotherapists in many countries, in which stimulation of central nervous system is to achieve the highest possible functional level
  Arms: PNF group
Other: manual therapy group — Manual therapy is used for an assessment and treatment of joint and soft tissues.
  The basic therapeutic tool is mobilisation. In the study joint mobilisation according to Kaltenborn-Evjenth Manual Therapy was used. The joint were mobilised with low velocity passive movements in the whole or end range. Spinal manipulation wasn't used. Liter Exelby reports that manual therapy with joints mobilisation was quite effective in improvement of functional movements and decreasing of pain.
  Arms: Manual therapy group

SUMMARY:
Abstract Objective: To compare effect of PNF therapy with manual therapy on pain, associated symptoms, range of motion and functioning in patients with cervical spine osteoarthritis.

Design: Parallel group, single-center, double-blinded randomized controlled trial.

Setting: Outpatient clinic in hospital KCRiO. Subject: Eligible patients were female adults with chronic pain of cervical spine due to osteoarthritis of vertebral body and intervertebral disc confirmed by X-ray.

Interventions: Group I (PNF group) was treated according to PNF concept, while Group II according to manual therapy (manual therapy group). Both groups received 10 days of treatment, 45 minutes each day.

Main measures: Primary outcomes measures were Oswestry scale and range of motion (ROM). Secondary outcomes measures were subjective evaluation of cervical pain according to VAS scale and associated symptoms (headache, vertigo, ROM of shoulder joints, balance). For each scale results were measured at baseline, after two weeks of intervention and after a three-month follow-up period without therapy.

Keywords: neck pain, PNF, manual therapy

DETAILED DESCRIPTION:
Degenerative changes of cervical spine contribute to pain and decreasing ROM. Cervical pain is the fourth common cause of disability in the United States and it has a significant socio-economic impact worldwide. Pain of cervical spine is one of the leading cause of decreasing quality of life and it requires more attention from medical service providers and researchers. Further sudies are urgently required to better understand prognostic factors and clinical course of neck pain especially in low-middle-income countries as well as ways how to prevent such ailments. Especially office workers run the risk of musculoskeletal system overload due to prolonged sitting position with office equipment not suited to their needs [4,5,6]. The annual incidence of neck pain in industrialised countries varies from 27% to 48% what generates high costs and becomes the key issue.

In 50-85% patients suffering from pain of cervical spine the symptoms don't resolve spontaneously and in 47% they may become chronic. Common cause of neck pain is: sedentery lifestyle, office work, difficulty sleeping, obesity, bad posture, depression, frequent use of a computer, female gender. Neck pain is common in office workers and it happens annual in 13-48% of them. As many as 42-69% experienced neck pain in last 12 months and in 34-49% they reported the beginning of neck pain during annual observation. Until now there are no clear conclusions concerning types of exercises to decrease pain and improve function of cervical spine in the proffesion mentioned. Neck pain often becomes chronic and it stays at least 6 months in 10% in man and 17% in women. Considering that neck pain is a problem for the general population it seems appropriate to indicate a treatment which will decrease pain effectively and that can improve functionig in daily living.

The goal of this study is to Compare the effect of PNF therapy with manual therapy in improving range of motion, decreasing pain, associated symptoms and improving ADLs in patients with cervical spine osteoarthtitis.

The parallel-group, single-centered, double-blind randomized experimental study was conducted in Cracow Rehabilitation and Orthopedic Centre in an outpatient clinic located in Aleja Modrzewiowa 22 in Poland. This medical facility has i.a. Accreditation Certificate, ISO Certificate. Written information was delivered to the Director of the Centre who obtained consent. The Bioethics Commission expressed a positive opinion on conducting the studies No. 71/KBL/OIL/2011 and follows the Declaration of Helsinki for ethical principles for medical research involving humans.

Patients admitted to rehabilitation in KCRiO were screened by Physical Medicine and Rehabilitation physician and on the basis of entry criteria they were qualified or excluded. All the patients involved were asked to sign a written informed consent for the participation in the study and filling in baseline assessments.The patients underwent rehabilitation program tailored for cervical osteoarthritis. One group received PNF treatment, the second one manual therapy. The patients were treated individually. Additionally both groups received physical modalities: laser therapy and TENS on cervical spine. Time of treatment was 2 weeks- 10 rehabilitation units 45 minutes each, once a day.

Treatment in the Ist group (PNF) included:

* neck patterns with a technique: Combination of Isotonics
* upper extremity patterns with a technique: Combination of Isotonics
* neck patterns with a technique: Hold-Relax
* scapula patterns with techniques: Stabilizing Reversals and Contract-Relax
* reeducation of postural control.

Treatment used in the IInd group (manual therapy) included:

* mobilisation of cervicothoracic junction
* cervical segmental mobilisation (flexion, extension, coupling movement)
* isometric exercises of cervical spine
* PIR (post-isometric muscle relaxation)
* traction of cervical spine
* received reeducation for postural control

Data was collected concerning age, BMI and type of work. After randomisation patients in both groups were blinded with regard to kind of received treatment and the study hipothesis. They received information who would be their physiotherapist. Data collecter was not involved in the trial. Observer collecting data couldn't enter the exercise room while patients were treated and couldn't be prezent during randomization. Contact between a person responsible for randomization process and data collector, as well as between caregivers and data collector was avoided; it was monitored by a Head of Physiotherapy Unit.

ELIGIBILITY:
Inclusion criteria:

* age 45-65,
* female gender,
* cervical pain due to osteoarthritis of vertebral body and intervertebral disc confirmed by X-ray,
* chronic pain lasting more than 13 weeks, verbal contact,
* intact cognitive functions and voluntary consent for the study.

Exclusion criteria

* birth or aquired deficits,
* cervical spine injury,
* osteoporosis,
* cervical spine instability,
* myelopathy,
* signs of nerve root compression of C1-C8, such as paresis, muscle loss, hyporeflexia, use of analgesics,
* anti-inflammatory drugs or myorelaxants.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Oswestry scale | Change from baseline Oswesstry scale at 2 weeks.
  Oswestry Disability Index (ODI) can be used for evaluation both cervical and lumbar spine. It is the most common method used for disability evaluation of patients with neck pain. It consits of questiones which evaluate how the pain limits activities. There are 10 questiones concerning ADLs.

SECONDARY OUTCOMES:
VAS scale | baseline, two weeks, 3 months
  One of the most commonly used scale for pain evaluation is Visual Analogue Scale (VAS). It is easy to use, it doesn't require any verbal or reading abilities and it's comprehensive enough. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left side.
assessment of the occurrence of vertigo, balance problems,nausea,limited ROM in shoulder joints | baseline, two weeks, 3 months
  There were closed questiones with yes or no answer
ROM evaluation | baseline, two weeks, 3 months
  ROM of cervical spine was evaluated with a measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Maicki, PhD, Principal Investigator — Jagiellonian University Colegium Medicum
Locations (1):
- Krakowskie Centrum Rehabilitacji i Ortopedii, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed Consent Form, will be made available
Supporting Information: Study Protocol, ICF
Time Frame: available
Access Criteria: on email request: tomasz.maicki@uj.edu.pl

REFERENCES:
- [Result] Nazari G, Bobos P, Billis E, MacDermid JC. Cervical flexor muscle training reduces pain, anxiety, and depression levels in patients with chronic neck pain by a clinically important amount: A prospective cohort study. Physiother Res Int. 2018 Jul;23(3):e1712. doi: 10.1002/pri.1712. Epub 2018 Mar 14. PMID 29536618
- [Result] Malik AA, Robinson S, Khan WS, Dillon B, Lovell ME. Assessment of Range of Movement, Pain and Disability Following a Whiplash Injury. Open Orthop J. 2017 Jul 19;11:541-545. doi: 10.2174/1874325001711010541. eCollection 2017. PMID 28839498
- [Result] Vincent K, Maigne JY, Fischhoff C, Lanlo O, Dagenais S. Systematic review of manual therapies for nonspecific neck pain. Joint Bone Spine. 2013 Oct;80(5):508-15. doi: 10.1016/j.jbspin.2012.10.006. Epub 2012 Nov 16. PMID 23165183
- [Result] de Koning CH, van den Heuvel SP, Staal JB, Smits-Engelsman BC, Hendriks EJ. Clinimetric evaluation of active range of motion measures in patients with non-specific neck pain: a systematic review. Eur Spine J. 2008 Jul;17(7):905-21. doi: 10.1007/s00586-008-0656-3. Epub 2008 Apr 22. PMID 18427843
- [Result] Ylinen J, Kautiainen H, Wiren K, Hakkinen A. Stretching exercises vs manual therapy in treatment of chronic neck pain: a randomized, controlled cross-over trial. J Rehabil Med. 2007 Mar;39(2):126-32. doi: 10.2340/16501977-0015. PMID 17351694
- [Result] Cunha AC, Burke TN, Franca FJ, Marques AP. Effect of global posture reeducation and of static stretching on pain, range of motion, and quality of life in women with chronic neck pain: a randomized clinical trial. Clinics (Sao Paulo). 2008 Dec;63(6):763-70. doi: 10.1590/s1807-59322008000600010. PMID 19060998
- [Result] Lluch E, Arguisuelas MD, Coloma PS, Palma F, Rey A, Falla D. Effects of deep cervical flexor training on pressure pain thresholds over myofascial trigger points in patients with chronic neck pain. J Manipulative Physiol Ther. 2013 Nov-Dec;36(9):604-11. doi: 10.1016/j.jmpt.2013.08.004. Epub 2013 Oct 21. PMID 24152997
- [Result] Falla D, O'Leary S, Farina D, Jull G. Association between intensity of pain and impairment in onset and activation of the deep cervical flexors in patients with persistent neck pain. Clin J Pain. 2011 May;27(4):309-14. doi: 10.1097/AJP.0b013e31820212cf. PMID 21178596
- [Result] Cleland JA, Childs JD, Fritz JM, Whitman JM, Eberhart SL. Development of a clinical prediction rule for guiding treatment of a subgroup of patients with neck pain: use of thoracic spine manipulation, exercise, and patient education. Phys Ther. 2007 Jan;87(1):9-23. doi: 10.2522/ptj.20060155. Epub 2006 Dec 1. PMID 17142640
- [Result] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741